CLINICAL TRIAL: NCT05176496
Title: Characterization and Treatment Pathways of Heavy Menstrual Bleeding (HMB)
Brief Title: A Study Called Champion-HMB to Learn More About Females With Heavy Menstrual Bleeding and Available Treatments to Enable Earlier Diagnosis and to Predict Courses of Treatment
Acronym: Champion-HMB
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22061
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Women with a continuous observation of 365 days after January 1st, 2000 and before December 31, 2020.
- Cohort 2: Women diagnosed with HMB.

SUMMARY:
This is an observational study in which patient data from the past of females with heavy menstrual bleeding (HMB) is studied.

• HMB describes menstrual periods with abnormally heavy or prolonged bleeding. Women concerned may not be able to maintain their usual activities during their period. Thus, HMB can reduce the quality of life and may lead to other medical problems. It is described that up to 30 of 100 women ask doctors for help concerning HMB during their fertile years. HMB is often not recognized and treated timely. In addition, there is little information about characteristics of women with HMB and real-world data on available treatments are missing.

Despite the availability of non-invasive therapeutic options, for some women with severe HMB, surgical treatments (also called invasive) may be needed that can lead to infertility.

* In this study researchers want to learn more about:
* the percentage of women diagnosed with HMB
* characteristics of these women like age at diagnosis or medical problems
* treatment pathways of women with HMB in usual care

Regarding treatment pathways, the researchers are especially interested in:

* the percentage of women who use different therapeutic options over time
* the percentage of women receiving invasive treatment for HMB after they received treatment as recommended by guidelines versus those not treated as recommended
* To do this, researchers will collect information from five observational healthcare databases. Data will be from the year 2000 up to 2020.
* Besides this data collection, no further tests or examinations are planned in this study.
* In future, this information shall help to identify women with HMB and to learn what information may predict if invasive treatment will be needed later on.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* Women may enter the cohort if they are between 11 and 55 years old and have a continuous observation of 365 days after the start of the observation period (from January 1, 2000 to December 31, 2020). Cohort entry events are limited to the earliest event per person.
* Entry events having no procedure occurrences of hysterectomy, starting anytime on or before cohort entry start date.
* Entry events having no condition occurrences of natural or iatrogenic menopause, starting anytime on or before cohort entry start date.

Cohort 2:

* Women between 11 and 55 years old with continuous observation of 365 days before event may enter the cohort when observing a condition occurrence of HMB for the first time in the person's history; starting between January 1st, 2000 and December 31st, 2020. Cohort entry events are limited to the earliest event per person.
* Entry events having no procedure occurrences of hysterectomy, starting anytime on or before cohort entry start date.
* Entry events having no condition occurrences of natural or iatrogenic menopause, starting anytime on or before cohort entry start date.
* Entry events having no condition occurrences of gynaecological bleeding other than HMB, starting anytime on or before cohort entry start date.

Cohort 3:

- The cohort entry events, index date, and exit events are identical to those defined for cohort 2. Inclusion criteria is as defined for cohort 2, plus adding entry events having no condition occurrences of underlying causes of HMB, listed in 9.2.4.2 Underlying causes of HMB and including polyps, adenomyosis, leiomyoma, malignancy and endometrial hyperplasia, coagulopathy or iatrogenic HMB, starting anytime before or after cohort entry start date.

Cohort 4:

- The cohort entry events, index date, and exit events are identical to those defined for cohort 2. Inclusion criteria is defined as for cohort 2, plus adding entry events having a prescription for LNGIUD or a procedure occurrence of LNG-IUD placement, starting anytime after cohort entry start date.

Cohort 5:

- The cohort entry events, index date, and exit events are identical to those defined for cohort 2. Inclusion criteria is defined as for cohort 2, plus adding entry events receiving a prescription for, or a procedure occurrence of a guideline treatment (e.g. a prescription for LNG-IUD or a procedure occurrence of LNG-IUD placement), starting anytime after cohort entry start date.

Cohort 6:

- The cohort entry events, index date, and exit events are identical to those defined for cohort 2. Inclusion criteria is defined as for cohort 2, plus adding entry events of not receiving a prescription for, or a procedure occurrence of a guideline treatment (e.g. a prescription for LNG-IUD or a procedure occurrence of LNG-IUD placement), starting anytime after cohort entry start date.

Cohort 7:

- The cohort entry events, index date, and exit events are identical to those defined for cohort 2. Inclusion criteria is defined as for cohort 2, plus adding entry events of receiving a diagnosis of endometrial hyperplasia, or endometrial or cervical cancer anytime time prior to or after cohort entry start date.

Exclusion Criteria:

- None.

Ages: 11 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes 11 to 55-year-old women diagnosed with HMB in France, Germany, UK and US from 2000 to 2020.
Sampling Method: Non-Probability Sample
Enrollment: 99999 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Incidence rates of women diagnosed with HMB per year | Retrospective analysis from 2000 to 2020
Incidence rates of women diagnosed with HMB over the entire study period | Retrospective analysis from 2000 to 2020
Proportion of women receiving a diagnosis of HMB over the entire study period | Retrospective analysis from 2000 to 2020
Patient characteristics of women with a diagnosis of HMB | Retrospective analysis from 2000 to 2020
  Characterize demographics, co-morbidities, co-medications, procedures.
Comorbidities of women with a diagnosis of HMB | Retrospective analysis from 2000 to 2020
Treatment pathways of multiple therapeutic options | Retrospective analysis from 2000 to 2020
Frequency of guideline-compliant treatment for HMB | Retrospective analysis from 2000 to 2020
Patient characteristics | Retrospective analysis from 2000 to 2020
  Characterise women with guideline-compliant versus non-guideline compliant treatment.
Frequency/incidence of future invasive treatment | Retrospective analysis from 2000 to 2020
  Characterise women with guideline-compliant versus non-guideline compliant treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.